CLINICAL TRIAL: NCT03107403
Title: Investigation of the Links Between Waking-life and Dream Content in the Case of the Death of a Close Relative
Brief Title: Dreams and Bereavement
Acronym: DreamDeath
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL17_0075; 2017-A00640-53 (Other: ID-RCB)
Record Dates: First submitted 2017-04-05; First posted 2017-04-11 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Healthy Subjects
Keywords: dreams bereavement; emotional; regulation; bereavement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy subjects (Experimental)
  Interventions: Behavioral: web form

INTERVENTIONS:
Behavioral: web form — The scale assessing the bereavement process is the one reported in Teissier 2010

SUMMARY:
The aim of the study is to investigate a possible role of dreaming in emotion regulation testing whether dreaming of a close relative recently deceased is correlated with a positive evolution of the bereavement process

ELIGIBILITY:
Inclusion Criteria:

* age > or = 18 years old
* the death of a close relative in the last 3 months

Exclusion Criteria:

- history of psychiatric and neurologic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2023-04-09 (Actual); Study Completion 2023-04-09 (Actual)

PRIMARY OUTCOMES:
Frequency of dreams related to the deceased will be correlated to the score at the scale assessing the bereavement process | Day 1
Frequency of dreams related to the deceased will be correlated to the score at the scale assessing the bereavement process | Day 90
Frequency of dreams related to the deceased will be correlated to the score at the scale assessing the bereavement process | Day 180
Frequency of dreams related to the deceased will be correlated to the score at the scale assessing the bereavement process | Day 270
Frequency of dreams related to the deceased will be correlated to the score at the scale assessing the bereavement process | Day 360

SECONDARY OUTCOMES:
Content of dreams related to the deceased will be correlated to the score at the scale assessing the bereavement process | Day 1
Content of dreams related to the deceased will be correlated to the score at the scale assessing the bereavement process | Day 90
Content of dreams related to the deceased will be correlated to the score at the scale assessing the bereavement process | Day 180
Content of dreams related to the deceased will be correlated to the score at the scale assessing the bereavement process | Day 270
Content of dreams related to the deceased will be correlated to the score at the scale assessing the bereavement process | Day 360

CONTACTS AND LOCATIONS:
Overall Officials: Alain Nicolas, MD, Principal Investigator — Hôpital le Vinatier/Inserm
Locations (1):
- Hospices Civils de Lyon Hôpital le Vinatier/Inserm, Bron, France

IPD SHARING:
Plan to Share IPD: No